CLINICAL TRIAL: NCT07123246
Title: "Effects of Rigid Tape in Patients With Chronic Achilles Tendinopathy"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Gonzalo Elias, Principal Investigator, University of Gran Rosario
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rigid Tape and Achilles Tendon
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Achilles Tendinopathy (AT)
Keywords: AT

STUDY DESIGN:
Intervention Model Description: clinical trial with experimental and placebo groups
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rigid Tape group (Experimental): All participants in this arm will use a rigid tape during 72 hours. The rigid tape will consist of applying a pre-tape (Hypafix) to the patient´s skin, followed by an inelastic tape (Strappal) over it. The purpose of applying a pre-tape is to protect the skin from injury and to promote adherence of the rigid tape. The Strappal tape will be applied in a circular motion over the Achilles tendon, above the point of maximum pain felt by the patient, with compression to generate a biomechanical effect. The outcomes will be assessed before, immediately after and at 72 hours.
  Interventions: Other: Rigid Tape
- Placebo Tape group (Placebo Comparator): The placebo tape will consist of applying a circular bandage to the mid-portion of the Achilles tendon. However, the pre-tape and a short piece of strappal will be applied without tension during its application, to avoid generating a biomechanical compression effect. The variables to be studied will be assessed before, immediately after, and 72 hours later.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Other: Rigid Tape — Inelastic rigid tape (Strappal) applied to discharge the Achilles tendon
  Arms: Rigid Tape group
Other: Placebo Control — A pre-tape and a short piece of rigid tape applied without tension.
  Arms: Placebo Tape group

SUMMARY:
The aim of this study will be to determine the clinical effects of rigid tape in patients with chronic MAT. The secondary outcomes will be to evaluate the immediate and short term pain, the height and pain during the vertical jump, the satisfaction of the use of the tape and the global rating of change (GROC) of the intervention. This study will be a double-blinded randomized clinical trial comprising a total sample size of 36 participants with MAT of both genders and aged between 18 and 50 years. Subjects will undergo a screening process by a sports medicine doctor by different diagnostic tests to identify those presenting a diagnosis of painful MAT and then, they will be randomized into either a group performing experimental rigid tape (G1), or a group performing placebo tape (G2). The study will assess the subjects immediate and short-term tendon pain following the tape application during running and vertical jump. Also the tape satisfaction and GROC will be assessed. The rigid tape will be applied in the central portion of the Achilles tendon. Primary and secondary outcomes will be measured at baseline, immediate after the application of the tape and 72 hours after. The GROC will only be assessed at the end of the treatment. All the evaluations will be performed by a blinded physiotherapist. The patient will also be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral or bilateral MAT
* Achilles pain > 3 months
* Age ranging between 18 to 50 years, both genders
* Read and speak Spanish well enough to provide informed consent and follow study instructions.
* Pain during running and jumping.

Exclusion Criteria:

* Any ankle or foot surgery
* History of Achilles rupture
* Heel pain in the last 3 months
* Systemic disorders/diseases
* Body mass index > 30kg/m2
* Self-report of pregnancy
* Pain < 2/100 of average pain on VAS
* VISA A score > 90 points

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change on pain intensity | At baseline, immediately and 72 hours after the intervention
  The Visual Analog Scale (VAS) will be used to assess pain intensity during running and jumping. This scale consists of a sequence of numbers from 0 (no pain) to 100 mm (most severe pain).

SECONDARY OUTCOMES:
Change on single leg vertical jump | At baseline, immediately and 72 hours after the intervention
  This test will assess the height in cm and power of a vertical jump using the My Jump app, validated by Gallardo-Fuentes in 2016. The instructions will be jumping as high as possible with hands on the subject's waist. Participants will perform 3 repetitions in a non-consecutive manner.
Change on feeling of comfort of the tape | Immediately and 72 hours after the intervention
  The satisfaction of the tape will be assessed by the Likert Scale. This rating scale measures the positive or negative response to the intervention. The format of this scale will be divided into five levels: "very uncomfortable", "uncomfortable", "normal", "comfortable", and "very comfortable".
Change in perception of improvement of the treatment | 72 hours after the intervention
  The Global Rating of Change (GROC) scale is a patient-reported outcome measure used to assess the subjective perception of change in a patient's condition following an intervention. It helps determine whether a patient's condition has improved, worsened, or remained the same since the start of treatment. The magnitude of this difference is recorded on an 11-point visual analog scale, starting from "0" (no change) as the midpoint, and presenting at its extremes "-5" (much worse) and "+5" (completely better).

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Silbernagel KG, Hanlon S, Sprague A. Current Clinical Concepts: Conservative Management of Achilles Tendinopathy. J Athl Train. 2020 May;55(5):438-447. doi: 10.4085/1062-6050-356-19. Epub 2020 Apr 8. PMID 32267723
- [Background] de Vries A, Zwerver J, Diercks R, Tak I, van Berkel S, van Cingel R, van der Worp H, van den Akker-Scheek I. Effect of patellar strap and sports tape on pain in patellar tendinopathy: A randomized controlled trial. Scand J Med Sci Sports. 2016 Oct;26(10):1217-24. doi: 10.1111/sms.12556. Epub 2015 Sep 17. PMID 26376953
- [Background] Dar G, Mei-Dan E. Immediate effect of infrapatellar strap on pain and jump height in patellar tendinopathy among young athletes. Prosthet Orthot Int. 2019 Feb;43(1):21-27. doi: 10.1177/0309364618791619. Epub 2018 Aug 13. PMID 30101673